CLINICAL TRIAL: NCT06353061
Title: Phase II Randomized Window of Opportunity Trial of Chemoradiotherapy Alone Versus Combination With Metformin in Locally Advanced Cervical Cancer
Brief Title: Chemoradiotherapy With or Without Metformin in Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACC-MET
Record Dates: First submitted 2024-03-10; First posted 2024-04-08 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer; Radiotherapy; Metformin; Hypoxia; PET/CT
Keywords: Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypoxia | interventions — Metformin; Radiotherapy; Drug Therapy; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group treated with metformin in combination with synchronous chemoradiotherapy (Experimental): After the group allocation is determined, patients in the experimental group will undergo CA-IX PET/CT scans. Subsequently, they will commence taking metformin at a dose of 850 mg per tablet, once daily, for three consecutive days. One week later, a second CA-IX PET/CT scan will be performed. Following this, synchronous chemoradiotherapy will be initiated, with patients taking metformin twice daily during the course of radiotherapy, at a dosage of one tablet per administration.
  Interventions: Drug: Metformin; Radiation: Radiotherapy; Drug: Chemotherapy; Diagnostic Test: PET/CT
- The group undergoing chemoradiotherapy alone. (Active Comparator): Patients in the control group will undergo the first CA-IX PET/CT scan after the group allocation. One week later, they will undergo the second PET/CT scan. Subsequently, they will commence synchronous chemoradiotherapy.
  Interventions: Radiation: Radiotherapy; Drug: Chemotherapy; Diagnostic Test: PET/CT

INTERVENTIONS:
Drug: Metformin — Patients randomized to the metformin group will start taking metformin within 1 day after group allocation. They will take one tablet of metformin (850 mg) once daily for three consecutive days. Subsequently, they will take metformin orally twice daily throughout the entire external and internal irradiation period, with each administration consisting of one tablet.
  Arms: The group treated with metformin in combination with synchronous chemoradiotherapy
Radiation: Radiotherapy — The study requires all subjects to sequentially undergo external beam radiotherapy (EBRT) and intracavitary brachytherapy (BT). All radiotherapy must be completed within 7-8 weeks after treatment initiation. The total prescribed dose EQD2 for EBRT combined with BT should be ≥80 Gy; for subjects with squamous carcinoma with lesions ≤4 cm, the HR-CTV D90 should be ≥80 Gy; for subjects with adenocarcinoma or lesions >4 cm, it is recommended that HR-CTV D90 should be ≥85 Gy. When the prescribed dose is limited by organs at risk (OAR), priority should be given to covering HR-CTV. The radiotherapy plan in this study is based on image guidance. Imaging scans can use MRI or CT, and the scanning area should extend at least 5 cm above and below the PTV.
Drug: Chemotherapy — The dosage of cisplatin is 40 mg/m2, administered once weekly during radiotherapy for a duration of 5 weeks. Prior to and following cisplatin administration, 1-2 liters of fluid should be given for adequate hydration. Treatment should continue until disease progression or intolerable toxicity occurs.
Diagnostic Test: PET/CT — Using 68Ga-NY104 as a small molecule targeted imaging agent for CA-IX, two CA-IX PET/CT scans will be conducted in patients: one upon enrollment and another one week after randomization.

SUMMARY:
This is a prospective, single-center, phase II, randomized, window-of-opportunity trial initiated by researchers. The research hypothesis is that metformin can improve the level of hypoxia in locally advanced cervical cancer and further improve progression-free survival. The study aims to compare the improvement of tumor hypoxia with synchronous chemoradiotherapy with or without metformin, using CA-IX PET/CT and radiation positioning spectral CT to evaluate tumor hypoxia, screening hypoxic patients for inclusion in the study, and comparing the effects of synchronous chemoradiotherapy with or without metformin on the degree of hypoxia and progression-free survival in the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-70 years old
2. Pathologically confirmed cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma
3. FIGO stage IB2-IVA
4. Baseline CT or MRI indicating tumor necrosis (clinical hypoxia)
5. Hemoglobin ≥90g/L (blood transfusions allowed); no prior chemotherapy
6. ECOG performance status 0-2
7. No severe hematopoietic dysfunction, and no significant cardiac, pulmonary, hepatic, renal dysfunction, or immune deficiency
8. Able to undergo PET/CT imaging
9. Feasible for gynecological examination and cervical biopsy
10. Not pregnant or breastfeeding

Exclusion Criteria:

1. Renal insufficiency with eGFR <45 ml‧min-1‧1.73 m-2, and acute conditions that may lead to renal impairment such as dehydration, severe infectious diseases, shock, etc.
2. Diagnosed diabetes mellitus or current use of metformin or any other antidiabetic medication.
3. Concurrent diseases that may lead to tissue hypoxia (especially acute or exacerbated chronic conditions), such as acute heart failure, pulmonary fibrosis, respiratory failure, recent myocardial infarction, or blood pressure monitoring showing less than 90/60 mmHg, SpO2 <90%.
4. Serum transaminases exceeding 3 times the upper limit of normal, liver failure, alcohol poisoning.
5. History of allergic reactions to compounds chemically or biologically similar to metformin.
6. Concurrent hypoglycemia, such as insulinoma, autoimmune hypoglycemia, or functional hypoglycemia, or fasting blood glucose persistently less than 2.8 mmol/L before enrollment.
7. Malnutrition, BMI <18.5.
8. Concurrent unhealed gastric ulcer, duodenal ulcer, ulcerative colitis, Crohn's disease, or recent episodes of severe abdominal pain, diarrhea, vomiting, etc.
9. Concurrent rectovaginal fistula, vesicovaginal fistula, uncontrolled vaginal bleeding, or those at risk of fistula.
10. Inability to undergo intracavitary radiotherapy as assessed by the investigator.
11. Human immunodeficiency virus (HIV) infection.
12. Severe underlying diseases that are untreatable.
13. History of other malignant tumors (excluding cured basal cell carcinoma of the skin) or previous pelvic radiotherapy.
14. Currently participating in other clinical trials or stopped participating in clinical trials less than 4 weeks ago.
15. Neurological or psychiatric abnormalities affecting cognitive function.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The degree to which metformin improves the hypoxic index measured by CAIX PET | 1week after randomization
  Using the uptake value parameter of CA-IX in PET/CT, comparing the changes in uptake values between the two scans as an indicator of improvement in hypoxia level

SECONDARY OUTCOMES:
Progression-free survival（PFS） | 2-year
  Progression-free survival is defined as the time from randomization to disease progression or death from any cause,whichever is first.
Changes in tumor volume during treatment | Baseline，1month and 2 months.
  Tumor volume will be measured via pelvic MRI.
Hematologic and gastrointestinal toxicities assessed by CTCAE v5.0 | Up to 3 months after treatment.
  Treatment-related toxicity reactions in both groups of patients will be evaluated during the treatment period, at the end of treatment, and three months after treatment completion
Quality of life assessed by QLQ-C30 | Up to 3 months after treatment
  Assessment of quality of life in both groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No